CLINICAL TRIAL: NCT03308214
Title: The Analysis of Factors Influencing the Apparent Volume of Distribution of Imipenem in Septic Shock Patients
Brief Title: The Analysis of Factors Influencing the Vd of Imipenem in Septic Shock Patients
Status: Completed | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Songqiao Liu, MD. PHD, Southeast University, China
Other Study IDs: 2017ZDSYLL073-P01
Record Dates: First submitted 2017-09-25; First posted 2017-10-12 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Septic Shock
Keywords: septic shock; imipenem; VD ;pharmacokinetics
MeSH Terms: conditions — Shock, Septic | interventions — Imipenem

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- septic shock: Patients with septic shock treat with Imipenem
  Interventions: Drug: Imipenem
- non-septic shock: Patients with infection but not septic shock treat with Imipenem
  Interventions: Drug: Imipenem

INTERVENTIONS:
Drug: Imipenem — Imipenem 1.0 q 8h

SUMMARY:
The study measures the plasma concentrations of imipenem in septic shock patients and non-septic shock patients and observes hypoalbuminemia and the impact of the severity of critical illness on Vd

DETAILED DESCRIPTION:
Severe sepsis and septic shock are major causes of mortality in intensive care unit(ICU) patients.Correct and adequate antibiotic coverage is essential but can be complex as a result of fluid resuscitation, hypoalbuminemia, organ dysfunction, the application of extracorporeal support modalities and the impact of critical illness on pharmacokinetics(PK).Such changes will significantly distort the normal anti-biotic PK profile, resulting in drug exposure that is markedly different from the 'healthy volunteer.'The apparent volume of distribution is one of important PK parameters.Vd determines the loading dose. This review article considers these issues in detail, summarizing the key changes in antibiotic Vd in the critically ill, and providing general suggestions how to optimization of antibiotic dosing to manage Vd challenges.50 patients who receives the theapy of imipenem are included in this study.Whether hypoalbuminemia, organ dysfunction, the application of extracorporeal support modalities and the impact of critical illness on Vd will be evaluted.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 years old and 80 years old;
2. Admitted to the ICU;
3. Patients diagnosed as septic shock requiring the therapy of imipenem(0.5g q6h or 1.0g q8h;

Exclusion Criteria:

1. Patient participated in another interventional trial before enrollment
2. Allergy, hypersensitivity or a serious reaction to imipenem;
3. Pregnancy.
4. patients with ECMO and(or)CRRT.
5. tumors.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: septic shock patients and non-septic shock patients with the therapy of imipenem in the ICU of Zhongda hospital
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-03-18 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
the apparent volume of distribution | Day1, Day 3, Day 7
  The imipenem plasma concentrations are measured at different time to calculate Vd

CONTACTS AND LOCATIONS:
Overall Officials: Songqiao Liu, PHD, Principal Investigator — Study Investigator
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang Y, Yang J, Xie J, Liu L, Liu S, Guo F, Qiu H, Yang Y. Association Between Pathophysiology and Volume of Distribution Among Patients With Sepsis or Septic Shock Treated With Imipenem: A Prospective Cohort Study. J Infect Dis. 2020 Mar 16;221(Suppl 2):S272-S278. doi: 10.1093/infdis/jiz651. PMID 32176787